CLINICAL TRIAL: NCT04179630
Title: A Phase 1, Single-center, Open Label, Parallel Group Study to Evaluate the Pharmacokinetics, Safety & Tolerability of a Single Dose of Aldafermin (NGM282) in Subjects With Impaired Renal Function
Brief Title: Study of Aldafermin (NGM282) in Participants With Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NGM Biopharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 282-RI-103
Record Dates: First submitted 2019-11-12; First posted 2019-11-27 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Impaired Renal Function
MeSH Terms: conditions — Renal Insufficiency | interventions — aldafermin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aldafermin (NGM282) (Experimental): Administered by subcutaneous injection
  Interventions: Biological: Aldafermin (NGM282)

INTERVENTIONS:
Biological: Aldafermin (NGM282) — Single 3 mg dose

SUMMARY:
This is a single-center evaluation of Aldafermin (NGM282) in an open-label, single-dose and parallel group study in participants with Impaired Renal Function.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of stable chronic kidney disease and eGFR, as assessed by the Modification of Diet in Renal Disease (MDRD) estimate:

  1. Mild renal impairment: eGFR 60-89 mL/min/1.73m²
  2. Moderate renal impairment: eGFR 30-59 mL/min/1.73m²
  3. Severe renal impairment: eGFR < 30 mL/min/1.73m²
* Healthy control subjects with normal renal function will be matched (age ± 10 years; sex, race, BMI ± 15%) to their respective subject in the impaired renal function groups and have eGFR ≥90 mL/min/1.73m . Healthy control subjects should have no systemic chronic disease.
* Males and Females age 18-75
* Body mass index (BMI) 25-40 kg/m²

Exclusion Criteria:

* Renal allograft recipients
* History of renal cell carcinoma or any history of metastatic disease involving the kidney
* End Stage Renal disease, requiring or not requiring dialysis
* Subject requiring or anticipated requirement of dialysis within 3 months of study entry
* Diagnosis of acute kidney injury/acute renal failure, or hospitalization for kidney related issue within 3 months of Screening
* Any renal disease or related condition actively being treated other than chronic kidney disease
* Any acute disease or condition being treated by medical therapy (prescription or over the counter) known to possibly impact renal function within 2 weeks of Screening
* History of treatment for a chronic condition with a medication that is known to have nephrotoxic potential, and after treatment, renal function/status has not been fully evaluated
* Uncontrolled hypertension
* Uncontrolled diabetes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-14 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of aldafermin (Day 1 through Day 4) | 12 Days
Area under the concentration-time curve from time zero extrapolated to infinity (AUC 0-infinity) of aldafermin (Day 1 through Day 4) | 12 Days

SECONDARY OUTCOMES:
Type and frequency of Adverse Events (Day 1 through Day 11) | 12 Days

CONTACTS AND LOCATIONS:
Overall Officials: NGM Study Director, Study Director — NGM Biopharmaceuticals
Locations (1):
- NGM Clinical Study Site, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided